CLINICAL TRIAL: NCT04576468
Title: The Use of Leucocyte Platelet Rich Fibrin (L- PRF) Covered Perforated Guided Tissue Membrane for Treatment of Periodontal Intrabony Defects (Randomized Clinical Trial)
Brief Title: The Use of Leucocyte Platelet Rich Fibrin (L- PRF) Covered Perforated Guided Tissue Membrane for Treatment of Periodontal Intrabony Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Mariam Samir, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDAS-RecIM011735
Record Dates: First submitted 2020-09-28; First posted 2020-10-06 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Periodontal Diseases
Keywords: perforated membrane; L-PRF; guided tissue regeneration; vertical defects; Intrabony defects
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: patients equally distributed into 4 groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- open flap debridement (Experimental): envelope full thickness flap reflection, removal of granulation tissue then suturing with simple loop sutures.
  Interventions: Procedure: Open flap debridement
- perforated membrane (PM) (Experimental): envelope full thickness flap reflection, removal of granulation tissue placing resorbable membrane after perforating it over the vertical defect then suturing with simple loop sutures.
  Interventions: Procedure: Open flap debridement; Procedure: perforated membrane
- leucocyte platelet rich fibrin (L-PRF) (Experimental): envelope full thickness flap reflection, removal of granulation tissue after withdrawal of blood and placing it in intraspin centrifuge , placing the resulting L-PRF in the defect then suturing with simple loop sutures.
  Interventions: Procedure: Open flap debridement; Procedure: leucocyte - platelet rich fibrin
- L-PRF + PM (Experimental): envelope full thickness flap reflection, removal of granulation tissue after withdrawal of blood and placing it in intraspin centrifuge , placing the resulting L-PRF covered by resorbable membrane after perforating it in the defect then suturing with simple loop sutures.
  Interventions: Procedure: Open flap debridement; Procedure: perforated membrane; Procedure: leucocyte - platelet rich fibrin

INTERVENTIONS:
Procedure: Open flap debridement — Surgical intevention
  Other Names: OFD
Procedure: perforated membrane — surgical intervention
  Other Names: perforated guided tissue membrane; regenerative surgery
  Arms: L-PRF + PM; perforated membrane (PM)
Procedure: leucocyte - platelet rich fibrin — surgical intervention
  Other Names: L-PRF; regenerative surgery
  Arms: L-PRF + PM; leucocyte platelet rich fibrin (L-PRF)

SUMMARY:
This study is the first to investigate the effect of leucocyte platelet rich fibrin (L-PRF) combined with perforated membrane in order to treat infrabony defects and assess their combined effect in clinical attachment level gain and filling of base of the defect (BD). The main hypothesis was that if the L-PRF act as a chemoattracttant for a higher number of periosteal derived periodontal cells (PDPCs) and gingival mesenchymal stem cells (GMSCs) encouraging their passage through the membrane perforations.

DETAILED DESCRIPTION:
A randomized (controlled) clinical trial which included forty sites with intrabony interproximal defects (2- or 3-wall) premolar/molar teeth assessed for clinical parameters. The four treatment modalities were randomly allocated by a predetermined computer generated randomization list (www.randomizer.org) into four equal groups; Group I (control group) open flap debridement (OFD): included intrabony defects treated by open flap debridement (OFD).Group II perforated membrane (PM): included intrabony defects treated by perforated membranes.Group III Leucocyte-platelet rich fibrin (L-PRF): included intrabony defects treated by leukocytes platelet rich fibrin (L-PRF). Group IV Leucocyte-platelet rich fibrin + perforated membrane (L-PRF + PM): included intrabony defects treated by Leucocyte platelet rich fibrin & perforated membranes.

ELIGIBILITY:
Inclusion Criteria:

* Both genders aged from 18- 60 years.
* Patients free from any systemic diseases that may contra-indicate periodontal surgery (Ahmed Y. Gamal et al., 2014).
* Two- or three-wall intrabony defects in premolar/molar teeth without furcation involvement, that are measured from the alveolar crest to the defect bottom in diagnostic periapical radiographs of ≥ 3 mm (Reynolds et al., 2015).
* Probing depth ≥ 5 mm and clinical attachment loss ≥ 4 mm at the site of intrabony defects 4 week after the phase one therapy (Ahmed Y. Gamal et al., 2014).
* Free from any periapical pathosis.
* Patients willing and able to return for multiple follow up visits and perform oral hygiene instructions.
* Absence of occlusal interference, mobility and open interproximal contact.
* Good fulfillment to plaque control instructions following initial therapy.

Exclusion Criteria:

* Smokers.
* Pregnant and breast feeding females.
* Periodontal surgical treatment in the previous 12 months at the involved sites. (A. Y. Gamal et al., 2016)
* Persistence of gingival inflammation after phase I therapy.
* Vulnerable groups as handicapped, mentally disabled, prisoners and orphans.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
clinical attachement level gain | 6 month
  measured using University of North Carolina Periodontal probe change from baseline at 6 month

SECONDARY OUTCOMES:
radiographic bone fill | 6 month
  measured using standardized periapical radiograph change from baseline at 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Y Gamal, Professor, Study Director — Faculty of dentistry - Ain shams University
Locations (1):
- Faculty of dentistry Ain shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No